CLINICAL TRIAL: NCT03029325
Title: Molecular and Genetic Analysis of Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Christopher Christiani, Elkan Blout Professor at Harvard TH Chan School of Public Health, Professor of Medicine Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 1999P-004935; 5P30CA006516-50 (NIH)
Record Dates: First submitted 2015-09-30; First posted 2017-01-24 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigators use a genome-wide approach within a case-control design to identify SNPs that show evidence of association with lung cancer risk and survival.

DETAILED DESCRIPTION:
Investigators also investigate how genetic variants may affect cancer treatment, at various stages of disease development, in order to determine prognostic and predictive factors for survival.

ELIGIBILITY:
Inclusion Criteria:

* healthy controls: participants without evidence of any cancer
* cases: pathology proven primary lung cancer

Exclusion Criteria:

* younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lung cancer cases and healthy controls are recruited from Massachusetts General Hospital patient population. Cases come from Thoracic Surgery or Cancer Center. Controls are usually spouses or friends of cases, or in some cases unrelated to a specific case.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 1993-06; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Survival among patients at different stages of lung cancer and treatment will be measured using questionnaires along with medical chart data to monitor treatment and disease progression | 20 years
  Study lung cancer development in a case control study. We will look at three separate outcome measures specified below

SECONDARY OUTCOMES:
Overall survival | 20 years
  Measurement from time of diagnosis to death will be obtained
Progression-free survival | 20 years
  Time of diagnosis to disease progression (measured by metastasis)
Treatment toxicities | 20 years
  Effects on ECOG and physical sequelae from treatment (radiation, chemotherapy and other treatment modalities will be analyzed)

CONTACTS AND LOCATIONS:
Overall Officials: David C Christiani, MD, Principal Investigator — Harvard TH Chan School of Public Health
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No